CLINICAL TRIAL: NCT05196581
Title: Randomized, Open-label Study to Evaluate the Efficacy of Breathox Device Inhalation Therapy in the Treatment of Acute Symptoms Associated With COVID-19 and in the Prevention of the Use of Health Resources in Patients With ≥ 18 Years Old
Brief Title: Efficacy of Breathox Device Inhalation Therapy in the Treatment of Acute Symptoms Associated With COVID-19 and in the Prevention of the Use of Health Resources
Acronym: BREATH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzana Erico Tanni Minamoto (Other)
Collaborators: Liita Care ApS (Industry)
Responsible Party: Sponsor-Investigator, Suzana Erico Tanni Minamoto, Clinical Professor, UPECLIN HC FM Botucatu Unesp
Organization: UPECLIN HC FM Botucatu Unesp (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BREA01
Record Dates: First submitted 2022-01-17; First posted 2022-01-19 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; sodium chloride
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No intervation (No Intervention): Thirty-four subjects receive no intervention.
- Experimental intervation one (Active Comparator): Thirty-three subjects receive dispersible NaCl powder, 8 mg per session per hour (one administration in each nostril and two oral inhalations), totaling 10 times a day, for ten days.
  Interventions: Drug: Dispersible NaCl powder 10 sessions
- Experimental intervation two (Active Comparator): Thirty-three subjects will receive dispersible NaCl powder, 8 mg per session (one administration in each nostril and two oral inhalations) every 3 hours, totaling 5 times a day, for ten days.
  Interventions: Drug: Dispersible NaCl powder 5 sessions

INTERVENTIONS:
Drug: Dispersible NaCl powder 10 sessions — Dispersible NaCl powder 10 sessions
  Other Names: Breathox
  Arms: Experimental intervation one
Drug: Dispersible NaCl powder 5 sessions — Dispersible NaCl powder 5 sessions
  Other Names: Breathox
  Arms: Experimental intervation two

SUMMARY:
SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2), the new coronavirus, causes a disease called COVID-19 that can trigger aggressive inflammatory responses. In this sense, in vitro intervention with high concentrations of sodium chloride has shown some favorable results in the inactivation of the disease Objective: to determine the effectiveness of inhaled sodium chloride therapy (BREATHOX®) in preventing the use of health resources in patients ≥ 18 years of age in 28 days compared to usual care. Method: Pilot, open randomized clinical trial study, including 100 patients with COVID-19 confirmed and symptomatic with up to 10 days of symptom onset. The included participants will be randomized according to a ratio of 1:1:1 into three groups: (Group 1) Standard of care + BREATHOX® one session (two oral inhalations and more nasal instillation in each nostril) every hour with a total of 10 sessions per day for 10 days; (Group 2) standard of care + BREATHOX® one session (two oral inhalations and more nasal instillation in each nostril) every three hours for a total of 5 sessions per day for 10 days; (Group 3) standard of care. After collecting the signed informed consent form, research participants will be evaluated on the tenth day of device use and re-evaluated on D28 for safety assessment. Recovery time for symptoms related to COVID-19 infection will be measured.

ELIGIBILITY:
Inclusion Criteria:

A. Adult males or females (≥ 18 years of age), not hospitalized, diagnosed with SARS-CoV-2 infection by oropharyngeal RT-PCR or swab antigen test, with mild symptoms of infection.

B. Symptomatic subjects must have at least 1 of the following symptoms at inclusion: fever or fever perceived for more than 24 hours, headache, sore throat, nasal obstruction, dry cough, fatigue, chest pain, or choking sensation (no associated respiratory distress ), myalgia, anosmia, ageusia or gastrointestinal symptoms within 10 days of onset;

C. Subjects with arterial pulse oximetry (SpO2) saturation ≥ 92% in room air at inclusion;

D. Participants with the following hematological and biochemical laboratory parameters obtained within 7 days before D0:

* Hemoglobin > 9.0 g/dL-1
* Absolute Neutrophil Count ≥ 1000 mm-³
* Platelets ≥ 100,000 mm-3
* Creatinine clearance ≥ 30 mL/min-1 by Cockcroft-Gault formula
* Rapid negative pregnancy test for women of childbearing age. and. Participants must understand, sign and date the voluntary written consent form at the visit prior to any protocol-specific procedure;

E. Participants must be able and willing to comply with study visits and procedures as per protocol.

Exclusion Criteria:

A. Moderate or severe acute respiratory failure, or requiring non-invasive ventilation or oxygen, or with SpO2 <92% or tachypnea (respiratory rate ≥30 breaths/minute);

B. Serious and uncontrolled preexisting organ insufficiency, which prevents participation in the study by the investigator's judgment;

C. Diagnosis of previous asthma using inhaled or oral corticosteroids in the last four weeks;

D. Previous use, in the last ten days of randomization, of inhaled, oral or intravenous corticosteroids; hydroxychloroquine and dewormers.

E. Previous diagnosis of chronic obstructive pulmonary disease, even when not using any inhaled medication;

F. Pregnant or lactating women;

G. Use of any investigational or unrecorded product within the 3 month period or the 5 half-lives period prior to the baseline period, whichever is longer;

H. Any condition that, in the investigator's opinion, could compromise the participant's safety or adherence to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of days of symptom clinic improvement | 10 days after treatment
  Number of days of symptom clinic improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No